CLINICAL TRIAL: NCT01993290
Title: Ultrasound-guided Brachial Plexus Block With the Single-penetration Multiple-injection-technique for Upper Extremity Surgery
Brief Title: USG Brachial Plexus Block for Upper Extremity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Borglum Neimann (Other)
Responsible Party: Sponsor-Investigator, Jens Borglum Neimann, Associate professor, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBH-PB; H-2-2012-055 (Other: The national committee on health research ethics)
Record Dates: First submitted 2013-06-10; First posted 2013-11-25 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Fracture at Wrist and/or Hand Level; Rupture of Tendon of Wrist and Hand; Injuries to the Wrist, Hand and Fingers (S60-S69); Ganglion Cysts; Carpal Tunnel Syndrome
MeSH Terms: conditions — Ganglion Cysts; Carpal Tunnel Syndrome | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- USG Supraclavicular block (Active Comparator): 20 ml of ropivacaine 0,75% is administered to brachial plexus at supraclavicular level.
  Interventions: Drug: Ropivacaine
- Lateral infraclavicular block (Active Comparator): 20 ml of ropivacaine 0,75 % is administered to brachialis plexus at lateral infraclavicular level
  Interventions: Drug: Ropivacaine
- USG Axillaris block (Active Comparator): 20 ml of ropivacaine 0,75% is administered to plexus brachialis at axillaris level
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 20 ml in total of 0,75% Ropivacaine is administered to each patient in all three arms.
  Other Names: Naropin

SUMMARY:
Ultrasound-guided (USG) brachial plexus (BP) block efficacy at the Supraclavicular (SCL), Lateral- Infraclavicular (LIC) and Axillary (AX) level: Randomized, observer-blinded study of the single-penetration multiple-injection-technique.

DETAILED DESCRIPTION:
The investigators will compare the BP block efficacy (for surgical anaesthesia) with the USG single-penetration multiple-injection-technique at the SCL, LIC and AX level for upper-extremity surgery (elbow, forearm, wrist, hand). The investigators want to investigate whether the single-penetration multiple-injection-technique would provide for safe surgical anaesthesia with lower volumes of local anaesthetics than has previously been described in a comparative study at the three different levels.

120 patients will prospectively be randomized to an USG BP block administered as a single-penetration multiple-injection-technique at one of three different levels: (1) SCL (2) LIC (3) AX. Ropivacaine 0.75% (20 mL) will be used for all blocks prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* American Society of Anaesthesiology class 1-3
* Patients undergoing upper extremity surgery

Exclusion Criteria:

* Inability to cooperate
* Inability to understand and talk danish
* Allergic to ropivacaine
* Infection at site of surgery
* Neurological dysfunction at site of surgery
* Severe coagulopathy
* Drug and alcohol abuse
* Patients, who can not get a nerve block due to technical difficulty
* Pregnancy or nursing
* Body mass index >35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Blockade performance time (seconds) | Time (seconds) from the time the ultrasound transducer is placed on the skin and until the needle is taken out of the body.

SECONDARY OUTCOMES:
Onset time of blockade (minutes) | Time from block completion to complete sensory and motor block is accomplished.
Number of needle passes | Number of times the direction of the needle changes while performing the block
Patient reported pain related to needle passes (Scale 0-2) | Pain related to block performance reported by the patient right after block completion
  0= no pain
  1. middle
  2. sever pain
Duration of time of block postoperatively (hours) | Patient reported the time off ending sensory and motory block

CONTACTS AND LOCATIONS:
Overall Officials: Mojgan Vazin, MD, Principal Investigator — Department of Anaesthesiology, Bispebjerg hospital
Locations (1):
- Department of anaesthesiology, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Koscielniak-Nielsen ZJ, Frederiksen BS, Rasmussen H, Hesselbjerg L. A comparison of ultrasound-guided supraclavicular and infraclavicular blocks for upper extremity surgery. Acta Anaesthesiol Scand. 2009 May;53(5):620-6. doi: 10.1111/j.1399-6576.2009.01909.x. PMID 19419356
- [Background] Mariano ER, Sandhu NS, Loland VJ, Bishop ML, Madison SJ, Abrams RA, Meunier MJ, Ferguson EJ, Ilfeld BM. A randomized comparison of infraclavicular and supraclavicular continuous peripheral nerve blocks for postoperative analgesia. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):26-31. doi: 10.1097/AAP.0b013e318203069b. PMID 21455085
- [Background] Tran DQ, Munoz L, Zaouter C, Russo G, Finlayson RJ. A prospective, randomized comparison between single- and double-injection, ultrasound-guided supraclavicular brachial plexus block. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):420-4. doi: 10.1097/AAP.0b013e3181ae733a. PMID 19920418